CLINICAL TRIAL: NCT02445261
Title: The Effects of Mobile Phone on Umbilical Artery Doppler and Fetal Cardiotogogrphy in Normal and Gowth Restricted Fetuses
Brief Title: Mobile Phone Effects on Umbilical Artery Doppler and Heart Rate Tracing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 133
Record Dates: First submitted 2015-05-11; First posted 2015-05-15 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Umbilical Artery Doppler; Fetal Heart Rate Tracing
Keywords: MOBILE PHONE ON AND IN AND; UMBILICAL ARTERY DOPPLER; FETAL CARDIOTOCOGRAPHY; GROWTH RESTRICTED FETUS; NORMAL GROWTH FETUS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- normal growth (Active Comparator): 120 woman with normal fetal growth will be subjected to 15 minutes CTG trace recording before using mobile phone and repeated while the phone is in the dialing mode for 10 minutes. Umbilical artery (UA) Doppler ultrasound will be done after the initial CTG trace and was repeated 5 minutes after hanging up the mobile phone. UA resistance indices, number of fetal kicks, the loss of acceleration and variability, and the appearance of decelerations were assessed
  Interventions: Radiation: mobile phone
- growth restricted group (Active Comparator): 70 woman with l growth restricted fetus will be subjected to 15 minutes CTG trace recording before using mobile phone and repeated while the phone is in the dialing mode for 10 minutes. Umbilical artery (UA) Doppler ultrasound will be done after the initial CTG trace and was repeated 5 minutes after hanging up the mobile phone. UA resistance indices, number of fetal kicks, the loss of acceleration and variability, and the appearance of decelerations
  Interventions: Radiation: mobile phone

INTERVENTIONS:
Radiation: mobile phone — Each woman was subjected to 15 minutes CTG trace recording before using mobile phone and repeated while the phone is in the dialing mode for 10 minutes. Umbilical artery (UA) Doppler ultrasound was done after the initial CTG trace and was repeated 5 minutes after hanging up the mobile phone.

SUMMARY:
Women were instructed not to use the mobile phones for 24 hours before carrying out the initial CTG trace and Doppler ultrasound. For each patient, initial 15 minutes CTG trace recording was done followed by umbilical artery Doppler ultrasound using high resolution ultrasound unit with 3-5 MHz transabdominal transducers (General Electric logic a500, logic a200 City country). Thereafter, the mobile phone (type, in the dialing mode, was put on the mother's abdomen for 10 minutes, concurrently with repeating the 15 minutes CTG trace. The umbilical artery Doppler was repeated 5 minutes after hanging up to avoid the interference with the Doppler machine. The umbilical artery Doppler ultrasound and the recorded fetal heart rate (FHR) strips before and after the mobile phone use were blindly analyzed with respect to umbilical artery resistance indices (RI) and CTG parameters in terms of number of fetal kicks, absence of beat to beat variability, loss of accelerations and the appearance of spontaneous decelerations.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 40 years pregnant between
* singleton fetus
* 32-38 weeks' gestation . They were classified into two groups. Group (A) included 120 women with normally growing fetuses. Group (B) included 70 women with growth-restricted fetuses.

Exclusion Criteria:

* presence of medical disorders or obstetric complications (in group A), anomalous fetus and non-reactive fetal CTG in initial CTG trace severe oligohydramnios

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2017-12-02 (Actual); Study Completion 2018-01-23 (Actual)

PRIMARY OUTCOMES:
umbilical artery doppler | 5 minutes after hanging up the mobile phone

SECONDARY OUTCOMES:
fetal heart rate tracing | 10 minutes after phone is in the dialing mode for

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Maged, Principal Investigator — Kasr Alainy medical school
Locations (2):
- Egypt (2):
  - Ahmed Maged, Cairo
  - Kasr Alainy medical school, Cairo